CLINICAL TRIAL: NCT03056391
Title: Effect of Paracetamol on Renal Function in Plasmodium Knowlesi Malaria: A Randomised Controlled Clinical Trial
Brief Title: Effect of Paracetamol on Renal Function in Plasmodium Knowlesi Malaria
Acronym: PACKNOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-16-356-29088
Record Dates: First submitted 2017-01-31; First posted 2017-02-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Malaria
Keywords: knowlesi malaria; paracetamol; renal function; haemolysis; oxidative stress
MeSH Terms: conditions — Malaria; Hemolysis | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Experimental): >50kg: Paracetamol 1gm PO/NG 6 hourly for 72 hours (maximum dose 4g/24h) plus IV artesunate or oral artemether/lumefantrine.
  <50kg: Paracetamol 12.5-15mg/kg/dose 6 hourly for 72 hours (maximum total dose 5doses/24hours;75mg/kg) plus IV artesunate or oral artemether/lumefantrine.
  Interventions: Drug: Paracetamol
- No Paracetamol (No Intervention): No Paracetamol plus IV artesunate or oral artemether/lumefantrine.
  If temperature >39.5°C, tepid sponging and mechanical antipyresis will be performed by research staff and/or relatives.

INTERVENTIONS:
Drug: Paracetamol — >50kg: Paracetamol 1gm PO/NG 6 hourly for 72 hours (maximum dose 4g/24h) plus IV artesunate or oral artemether/lumefantrine.
  <50kg: Paracetamol 12.5-15mg/kg/dose 6 hourly for 72 hours (maximum total dose 5doses/24hours;75mg/kg) plus IV artesunate or oral artemether/lumefantrine.
  Other Names: acetaminophen
  Arms: Paracetamol

SUMMARY:
Acute kidney injury is a common complication of severe Plasmodium knowlesi malaria, and an important contributor to mortality.

The exact pathogenic mechanisms of AKI in knowlesi malaria are not known, however it is hypothesised that haemolysis of red blood cells and subsequent release of cell-free haemoglobin leads to oxidative stress and lipid peroxidation in the renal tubules.

A novel mechanism of paracetamol was recently demonstrated, showing that paracetamol acts as a potent inhibitor of hemoprotein-catalyzed lipid peroxidation. In a proof of concept trial, paracetamol at therapeutic levels was shown to significantly decrease oxidative kidney injury and improve renal function by inhibiting the hemoprotein-catalyzed lipid peroxidation in a rat model of rhabdomyolysis-induced renal injury.

The investigators hypothesize that this novel inhibitory mechanism of paracetamol may provide renal protection in adults with knowlesi malaria by reducing the hemoprotein-induced lipid peroxidation that occurs in haemolytic conditions. As there is currently no consensus that exists concerning adequate medical treatment for severe malaria complicated by intravascular haemolysis and AKI, the potential application of paracetamol would be of benefit, especially as it is safe and widely available.

DETAILED DESCRIPTION:
Plasmodium knowlesi is the most common cause of malaria, and malaria deaths, in Sabah, Malaysia. Acute kidney injury (AKI) is a common feature of severe knowlesi malaria; however the mechanisms of AKI in knowlesi malaria are unknown. In falciparum malaria, recent evidence suggests that oxidative stress from haemolysis-related cell-free haemoglobin (CFHb) may contribute to pathogenesis of AKI.

Cell-free haemoglobin and oxidative stress: CFHb is released during intravascular haemolysis, and when exceeding the binding capacity of plasma haptoglobin, is filtered by the glomeruli and enters the renal tubules. CFHb is pathogenic as the ferrous heme can be oxidized to the ferric state, conferring peroxidase activity to the hemoglobin. Consequently, the hemoglobin can reduce hydroperoxides, such as hydrogen peroxide (H2O2) and lipid hydroperoxides, which generate the ferryl state of heme (FeIV=O) and a protein radical. The ferryl heme and protein radical can then generate lipid radicals by oxidation of free and phospholipid-esterified unsaturated fatty acids. The arachidonic side chains of membrane phospholipids are particularly vulnerable to this free radical-mediated damage in the complex cascade of lipid oxidation leading to the generation of F2-isoprostanes (F2-IsoPs) and isofurans (IsoFs). F2-IsoPs and IsFs are increased in severe falciparum malaria, and have been shown to induce vasoconstriction associated with renal injury in other haemolytic conditions including rhabdomyolysis, sepsis and post-operatively.

Paracetamol and oxidative stress: A novel mechanism of paracetamol was recently demonstrated, showing that paracetamol acts as a potent inhibitor of hemoprotein-catalyzed lipid peroxidation by reducing ferryl heme to its less toxic ferric state and quenching globin radicals. In a proof of concept trial, paracetamol at therapeutic levels was shown to significantly decrease oxidative kidney injury and improve renal function by inhibiting the hemoprotein-catalyzed lipid peroxidation in a rat model of rhabdomyolysis-induced renal injury. In a retrospective study of patients with sepsis, receiving paracetamol in the setting of raised CFHb was associated with reduced lipid peroxidation, and reduced risk of death. More recently, in a randomized placebo-controlled trial, paracetamol was associated with a reduction in F2-IsoPs and improved renal function in adults with sepsis and detectable CFHb.

Rationale: The investigators hypothesize that paracetamol may provide renal protection in patients with severe knowlesi malaria by reducing the hemoprotein-induced lipid peroxidation that occurs in haemolytic conditions. As there is currently no consensus that exists concerning adequate medical treatment for severe malaria complicated by intravascular haemolysis and AKI, the potential application of paracetamol would be of great benefit, especially as it is safe and widely available.

Proposed activities: The main activity proposed is a randomised, open label, controlled trial of regularly-dosed paracetamol, versus no paracetamol, in patients with knowlesi malaria, to assess the effect of paracetamol on renal function and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 5 years
2. Presence of P. knowlesi malaria, confirmed by positive blood smear with asexual forms of P. knowlesi.
3. Temperature >38C on admission or fever during the preceding 48 hours
4. Enrolled within 18 hours of commencing antimalarial treatment
5. Written informed consent from patient or attending relative able to and willing to give informed consent. Consent form and information sheets will be translated into Malay and copies provided to the patient.

Exclusion Criteria:

1. Patient or relatives unable or unwilling to give informed consent
2. Contraindication or allergy to paracetamol or artesunate therapy
3. Known cirrhosis, or >6 standard alcoholic drinks/day
4. Pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Effect of Paracetamol on kidney function | 72 hours
  Change in creatinine concentration (umol/L) at 72 hours from enrolment in patients receiving regularly-dosed paracetamol compared to those not receiving regular paracetamol, stratified by the level of intravascular haemolysis (cell-free haemoglobin).

SECONDARY OUTCOMES:
Longitudinal change in creatinine | 72 hours
  Longitudinal change in creatinine, as measured by the area under the creatinine-time curve, with creatinine measured 12 hourly from enrolment to 72 hours; and the effect of enrolment cell-free haemoglobin on longitudinal change in creatinine
Change in creatinine in severe malaria | 72 hours
  Change in creatinine at 72 hours and longitudinal change in creatinine over 72 hours, including the effect of enrolment CFHb, in patients with severe knowlesi malaria.
Development of AKI | 72 hours
  Development of AKI over 72 hours: i) an absolute increase in serum creatinine of >26.5 umol/L from enrolment creatinine; ii) a percentage increase in serum creatinine of >50% from enrolment; iii) post-enrolment onset of oliguria of less than 0.5ml/kg/hour for more than 6 hours; iv) 24 hour urine output of <400ml after rehydration and urinary obstruction excluded. AKI on enrolment will also be described by the Kidney Disease Improving Global Outcomes (KDIGO) criteria (with baseline creatinine estimated using the MDRD equation).
Duration of AKI | 28 days
  Length of time elapsed until serum creatinine returns to normal (estimated using MDRD equation) in the absence of renal replacement therapy in those with AKI on enrolment and those that develop AKI after enrolment.
Longitudinal changes in haemolysis: plasma cell-free haemoglobin | 72 hours
  Longitudinal changes in plasma cell-free haemoglobin over 72 hours.
Longitudinal changes in haemolysis: plasma cell-free haem | 72 hours
  Longitudinal changes in plasma cell-free haem over 72 hours.
Longitudinal changes in haemolysis: haem-to-protein cross-links | 72 hours
  Longitudinal changes in haem-to-protein cross-links over 72 hours.
Longitudinal changes in markers of oxidative stress: F2-IsoP | 72 hours
  Longitudinal changes in plasma F2-isoprostanes [F2-IsoP] over 72 hours.
Longitudinal changes in markers of oxidative stress: IsoF | 72 hours
  Longitudinal changes in plasma isofurans [IsoF]) over 72 hours.
Longitudinal changes in F2-IsoPs according to G6PD enzyme activity | 72 hours
  Longitudinal changes in F2-IsoPs according to G6PD enzyme activity, assessed qualitatively by fluorescent spot test.
Longitudinal changes in IsoFs according to G6PD enzyme activity | 72 hours
  Longitudinal changes in IsoFs and CFHb according to G6PD enzyme activity, assessed qualitatively by fluorescent spot test.
Longitudinal changes in CFHb according to G6PD enzyme activity | 72 hours
  Longitudinal changes in CFHb according to G6PD enzyme activity, assessed qualitatively by fluorescent spot test.
Longitudinal changes in F2-IsoPs according to G6PD genotype | 72 hours
  Longitudinal changes in F2-IsoPs according to G6PD genotype
Longitudinal changes in IsoFs according to G6PD genotype | 72 hours
  Longitudinal changes in IsoFs according to G6PD genotype
Longitudinal changes in CFHb according to G6PD genotype | 72 hours
  Longitudinal changes in CFHb according to G6PD genotype
Population pharmacokinetics of paracetamol: Cmax | 72 hours
  Peak plasma concentration (Cmax)
Population pharmacokinetics of paracetamol: Tmax | 72 hours
  Time to peak plasma concentration (Tmax)
Population pharmacokinetics of paracetamol: AUC | 72 hours
  Area under the plasma drug concentration-time curve (AUC)
Population pharmacodynamics of paracetamol | 72 hours
  Paracetamol dose-response curve
Fever clearance time | 72 hours
  Defined as the time taken for the aural temperature to fall below 37.5°C, and the time taken for the temperature to fall below 37.5°C and remain there for at least 24hours
Fever duration | 72 hours
  Defined as the duration in hours that an individual's temperature is above 37.5°C
Area above the fever versus time curve (AUC-T°) | 72 hours
  Area above the 37.5°C temperature versus time curve (AUC-T°) within first 24 hours of treatment.
Parasite clearance time (hours) | 72 hours
  Parasite clearance time, defined as (i) the time from commencement of antimalarial treatment to the first of 2 consecutive negative blood films, with blood films assessed by microscopy every 6 hours for the presence of asexual parasitaemia, and (ii) the linear portion of the slope of the log-parasitemia versus time relationship.
Blood and urine biomarkers of pre-renal and renal injury | 72 hours
  Neutrophil gelatinase-associated lipocalcin (NGAL), kidney injury molecule (KIM), urinalysis, urine microscopy, urine electrolytes, and urine creatinine.
Longitudinal urine colour | 72 hours
  Longitudinal urine colour (assessed by standardized urine colour charts). The proportion of patients with enrolment urine pH less than 6 together with a urine color of 6 or greater who develop AKI will be compared between groups.
Longitudinal urine pH | 72 hours
  Longitudinal urinalysis dipstick test-strip: urine pH. The proportion of patients with enrolment urine pH less than 6 together with a urine color of 6 or greater who develop AKI will be compared between groups.
Longitudinal urine specific gravity | 72 hours
  Longitudinal urinalysis dipstick test-strip: urine specific gravity
Longitudinal urine haemoglobin | 72 hours
  Longitudinal urinalysis dipstick test-strip: urine haemoglobin
Change in creatinine (umol/L) between therapeutic concentrations of paracetamol vs those with absent or low. | 72 hours
  Change in creatinine at 72 hours and longitudinal change in creatinine over 72 hours in patients with therapeutic concentrations of paracetamol, compared to patients with absent or low concentrations of paracetamol
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 days
  Reporting of any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with paracetamol administration
Longitudinal red cell deformability | 72 hours
  Longitudinal red cell deformability, as measured by laser-assisted optical rotational red cell analyser (LORCA) elongation index.
Longitudinal changes in markers of endothelial dysfunction | 72 hours
  Longitudinal changes in markers of weibel palade body exocytosis including angiopoietin-2

CONTACTS AND LOCATIONS:
Overall Officials: Giri M Rajahram, MD, Principal Investigator — Clinical Research Center, Queen Elizabeth Hospital, Kota Kinabalu, Sabah, Malaysia; Bridget Barber, MBBS, Study Director — Menzies School of Health Research; Nicholas Anstey, PhD, Study Director — Menzies School of Health Research; Matthew Grigg, MBBS, Study Director — Menzies School of Health Research; Timothy William, MBBS, Study Director — Jesselton Medical Centre; Jayaram Menon, MBBS, Study Director — Ministry of Health, Malaysia; Tsin Yeo, MBBS, Study Director — Menzies School of Health Research; Katherine Plewes, MD, Study Director — Mahidol Oxford Tropical Medicine Research Unit, Bangkok, Thailand; Arjen Dondorp, MD, Study Director — Mahidol Oxford Tropical Medicine Research Unit, Bangkok, Thailand; Daniel Cooper, MBChB, Study Director — Menzies School of Health Research
Locations (4):
- Malaysia (4):
  - Keningau District Hospital, Keningau, Sabah
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Kota Marudu District Hospital, Kota Marudu, Sabah
  - Ranau District Hospital, Ranau, Sabah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longley RJ, Grigg MJ, Schoffer K, Obadia T, Hyslop S, Piera KA, Nekkab N, Mazhari R, Takashima E, Tsuboi T, Harbers M, Tetteh K, Drakeley C, Chitnis CE, Healer J, Tham WH, Sattabongkot J, White MT, Cooper DJ, Rajahram GS, Barber BE, William T, Anstey NM, Mueller I. Plasmodium vivax malaria serological exposure markers: Assessing the degree and implications of cross-reactivity with P. knowlesi. Cell Rep Med. 2022 Jun 21;3(6):100662. doi: 10.1016/j.xcrm.2022.100662. PMID 35732155
- [Derived] Cooper DJ, Grigg MJ, Plewes K, Rajahram GS, Piera KA, William T, Menon J, Koleth G, Edstein MD, Birrell GW, Wattanakul T, Tarning J, Patel A, Wen Yeo T, Dondorp AM, Anstey NM, Barber BE. The Effect of Regularly Dosed Acetaminophen vs No Acetaminophen on Renal Function in Plasmodium knowlesi Malaria (PACKNOW): A Randomized, Controlled Trial. Clin Infect Dis. 2022 Oct 12;75(8):1379-1388. doi: 10.1093/cid/ciac152. PMID 35180298
- [Derived] Cooper DJ, Plewes K, Grigg MJ, Rajahram GS, Piera KA, William T, Chatfield MD, Yeo TW, Dondorp AM, Anstey NM, Barber BE. The effect of regularly dosed paracetamol versus no paracetamol on renal function in Plasmodium knowlesi malaria (PACKNOW): study protocol for a randomised controlled trial. Trials. 2018 Apr 24;19(1):250. doi: 10.1186/s13063-018-2600-0. PMID 29690924